CLINICAL TRIAL: NCT02815514
Title: Deutsches TAVI-Register
Brief Title: German TAVI-Register
Acronym: TAVI
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: TAVI
Record Dates: First submitted 2011-03-22; First posted 2016-06-28 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2016-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: aortic valve stenosis; aortic valve insufficiency; transapical aortic valve implantation; aortic valve replacement; percutaneous aortic valve replacement; aortic valve valvuloplasty
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic valve procedures: 1. percutaneous transfemoral aortic valve implantation
  2. percutaneous transapical aortic valve implantation
  3. percutaneous transaortic aortic valve implantation
  4. aortic valve valvuloplasty
  5. surgical aortic valve replacement
  6. conservative treatment

SUMMARY:
The TAVI - Register is a Germany-wide scientific elevation in which data about the aortic valve treatment and the therapeutic consequences are documented.

DETAILED DESCRIPTION:
Documentation of all consecutive patients of the participating centers with significant aortic stenosis, undergoing one of the following therapies:

1. Percutaneous transfemoral aortic valve replacement
2. Percutaneous aortic valve replacement transapical
3. Percutaneous aortic valve replacement transaortic
4. Aortic valve balloon valvuloplasty
5. Surgical aortic valve replacement
6. Conservative treatment

   * Documentation of the indications, procedural results and clinical short-and long-term results of the above therapies
   * Documentation of operational risk and quality of life
   * Documentation of the technical implementation of the procedure and success of the intervention and of hospital reinterventions
   * Documentation of hospital mortality, nonfatal major complications (stroke, TIA, myocardial infarction, dialysis, vascular complications, bleeding, neuropsychological status)
   * Documentation of discharge medication and the length of hospital stay
   * Documentation of the serious long-term complications, including mortality, stroke, TIA, myocardial infarction, dialysis, the reintervention and quality of life and of drug therapy within 30 days, 1 year, 3 years and 5 years.

ELIGIBILITY:
Inclusion Criteria:

patients with aortic stenosis (degree III) who received one of the following therapies:

* transapical operative aortic valve implantation
* operative aortic valve implantation
* percutaneous aortic valve implantation
* balloon valvuloplasty

Exclusion Criteria:

* missing signed informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with significant aortic valve stenosis, treated with aortic valve procedures.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 5 years

SECONDARY OUTCOMES:
Short- and long-term results of the documented therapies | 5 years
  Documentation of procedural results and clinical short-and long-term results of the documented therapies
Details on operational risk | up to four weeks
  Data are not recorded at a fixed day, but are collected during the initial hospital stay and are submitted when the patient leaves the hospital.
Details of performed procedures | up to four weeks
  Documentation of the indications, the technical implementation of the procedures and success of the intervention and of possible hospital reinterventions.
  Data are not recorded at a fixed day, but are collected during the initial hospital stay and are submitted when the patient leaves the hospital.
Complications during hospital stay | up to four weeks
  Documentation of hospital mortality, nonfatal major complications (stroke, TIA, myocardial infarction, dialysis, vascular complications, bleeding, neuropsychological status).
  Data are not recorded at a fixed day, but are collected during the initial hospital stay and are submitted when the patient leaves the hospital.
Details of hospital stay | up to four weeks
  Documentation of e.g. drug treatment, discharge medication and the length of hospital stay.
  Data are not recorded at a fixed day, but are collected during the initial hospital stay and are submitted when the patient leaves the hospital.
Serious long-term complications | 5 years
  Documentation of the serious long-term complications, including mortality, stroke, TIA, myocardial infarction, dialysis and reinterventions
Quality of life | 5 years
Drug treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Senges, MD, Principal Investigator — Stiftung Insitut fuer Herzinfarktforschung
Locations (1):
- Institut fur Herzinfarktforschung Ludwigshafen, Ludwigshafen, RPF, Germany

IPD SHARING:
Plan to Share IPD: No